CLINICAL TRIAL: NCT06172127
Title: A Multicenter, Open-Label, Single-Arm, Phase II Trial Exploring the Maintenance of Trastuzumab and Pertuzumab Following Trastuzumab Deruxtecan as Induction Treatment for HER2+ Unresectable Locally Recurrent or Metastatic Breast Cancer
Brief Title: PHESGO Maintenance After T-DXd Short Induction for HER2+ Unresectable Locally Recurrent or Metastatic Breast Cancer
Acronym: DEMETHER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDOPP562; 2023-507306-13-00 (Other: EU CT number); MO44772 (Other: F. Hoffmann-La Roche Ltd)
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2+ Breast Cancer; Unresectable Locally Advanced Breast Cancer; Metastatic Breast Cancer; PHESGO; Pertuzumab and Trastuzumab; T-DXd
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Injections

STUDY DESIGN:
Intervention Model Description: Single arm, non-comparative, phase 2 short induction treatment phase followed by maintenance treatment phase clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- T-DXd induction treatment phase followed by PHESGO maintenance treatment phase (Experimental): All patients will receive a 6-cycle induction phase with T-DXd 5.4 mg/kg body weight administered as an intravenous (IV) infusion on day 1 (D1) of each 21-day cycle (Q3W).
  Participants may continue with PHESGO if T-DXd is discontinued prematurely due to unacceptable toxicity prior to disease progression and following recovering to Grade ≤ 1 toxicity, to Grade 0 in case of ILD/pneumonitis, or to Grade 2 for alopecia/other toxicities not considered a safety risk. If any T-DXd unacceptable toxicity occurs during the first 6 cycles of induction phase with T-DXd, participants may receive taxane-based chemotherapy concomitantly with PHESGO treatment at the discretion of the investigator.
  During the maintenance phase, all participants will receive PHESGO with a loading dose of 1200 mg pertuzumab/600 mg trastuzumab as a SC injection for 8 minutes on D1 of the first 21-day cycle, and with a maintenance dose of 600 mg pertuzumab/600 mg trastuzumab as a SC Q3W.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Phesgo 1,200 MG / 600 MG / 30,000 UNT Per 15 ML Injection; Drug: Phesgo 600 MG / 600 MG / 20,000 UNT in 10 mL Injection

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — 10 mL type 1 amber borosilicate glass vial sealed with a fluoro-resin laminated butyl rubber stopper, and a polypropylene/aluminium yellow flip-off crimp cap. One vial of powder for concentrate for solution for IV infusion contains 100 mg of T-DXd. The drug product also contains L-histidine, L-histidine hydrochloride monohydrate, Sucrose, and Polysorbate 80.
  Other Names: T-DXd
Drug: Phesgo 1,200 MG / 600 MG / 30,000 UNT Per 15 ML Injection — 20 mL type I borosilicate glass vial tapered with fluororesin-laminated rubber stopper sealed with aluminum and covered by a cool green plastic flip-off cap, containing 15 mL solution of 1200 mg of pertuzumab and 600 mg of trastuzumab.
  Other Names: PHESGO; Pertuzumab-Trastuzumab FDC SC
Drug: Phesgo 600 MG / 600 MG / 20,000 UNT in 10 mL Injection — 15 mL type I borosilicate glass vial tapered with fluororesin-laminated rubber stopper sealed with aluminum and covered by a cool green plastic flip-off cap, containing 10 mL solution of 600 mg of pertuzumab and 600 mg of trastuzumab.
  Other Names: PHESGO; Pertuzumab-Trastuzumab FDC SC

SUMMARY:
DEMETHER is a phase II trial exploring the maintenance of trastuzumab and pertuzumab fixed dose combination (FDC) for subcutaneous administration (SC, PHESGO) following trastuzumab deruxtecan (T-DXd) as induction treatment for HER2-positive unresectable locally recurrent or metastatic breast cancer (MBC) patients.

DETAILED DESCRIPTION:
DEMETHER is an international, multicenter, open-label, single arm phase II clinical trial designed to evaluate the efficacy of a 6-cycle induction phase with T-DXd treatment followed by a maintenance phase with PHESGO treatment in patients with HER2-positive unresectable locally recurrent or MBC.

Upon meeting all selection criteria, a total of 165 participants will be enrolled. Participants with no prior chemotherapy or HER2-targeted therapy for advanced or MBC (one prior line of endocrine therapy is allowed for MBC) will be eligible. Participants who have received neoadjuvant or adjuvant chemotherapy will be eligible, with a DFI from completion of systemic chemotherapy to advanced or metastatic diagnosis of > 12 months.

Patients will continue study treatment until end of treatment (EoT) defined as the date of disease progression, death, discontinuation from the study treatment for any other reason, or up to 3 years (36 months) after T-DXd initiation, whichever occurs first. After discontinuation, all participants will undergo a safety visit at 28 (± 7 days) days after last treatment dose in order to follow up toxicities and changes in concomitant medication. Patients discontinuing the study treatment at any time will enter a post-treatment follow-up period during which survival and subsequent anticancer therapy information will be collected every 3 months (± 7 days) from the safety visit until death, lost to follow-up, elective withdrawal from the study, or the end of study (EoS), whichever occurs first.

The main objectives of DEMETHER study are to determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of progression-free survival (PFS) rate at 1 year and overall survival (OS) rate at 3 years.

End of study (EoS) is defined as the last data collection point at the last participant's safety visit and occur 36 months + 28 days (± 7 days) after the last patient included in the study initiates T-DXd treatment, unless premature termination of the study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet ALL the following criteria:

1. Patient must be capable to understand the purpose of the study and have signed written informed consent form (ICF) prior to beginning specific protocol procedures.
2. Male or female patients ≥ 18 years of age at the time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
4. Life expectancy of ≥ 12 weeks at screening.
5. Evidence of HER2-overexpressing tumor status confirmed by any MEDSIR's designated central lab or patient has a pathology report confirming HER2-overexpression by local testing, preferably on the most recent available metastatic sample. In the latest case, tumor tissue or blood must be sent to any MEDSIR's designated central lab for confirmation of HER2 status. Analysis of the primary tumor sample will be accepted if the metastatic tissue is inaccessible.
6. Must have known estrogen receptor (ER) and progesterone receptor (PgR) status locally determined prior to study entry.
7. Unresectable locally recurrent or MBC documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
8. Evaluable disease as per Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v.1.1) criteria.
9. Willingness and ability to provide the most recently available formalin-fixed paraffin-embedded (FFPE) tumor tissue blocks at the time of the inclusion (mandatory). If archival tissue is not available, a newly obtained baseline biopsy of an accessible tumor lesion is required prior to start of study treatment.
10. No prior chemotherapy and/or HER2-targeted therapy for advanced disease (one prior line of endocrine therapy is allowed for MBC).
11. May have received adjuvant or neoadjuvant chemotherapy and/or HER2-targeted therapy before study treatment initiation, with a disease-free interval (DFI) from completion of the systemic treatment (excluding hormonal therapy) to metastatic diagnosis of at least 12 months.
12. Adequate hematologic and organ function, defined by the following:

    1. Hematological (without platelet, red blood cell transfusion, and/or granulocyte colony-stimulating factor support within seven days before first study treatment dose): White blood cell (WBC) count > 3.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100.0 x 109/L, and hemoglobin (Hb) ≥ 9.0 g/dL.
    2. Hepatic: Serum albumin ≥ 2.5 g/dL; total bilirubin ≤ 1.5 times the upper limit of normal (x ULN) (≤ 3 x ULN in patients with known history of Gilbert's disease); alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5 × ULN in patients with liver and/or bone metastases); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 1.5 x ULN (≤ 3 x ULN in patients with liver metastases).
    3. Renal: Creatinine clearance ≥ 50 mL/min as determined by Cockcroft Gault (using actual body weight).
    4. Coagulation: International normalized ratio or prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN.
13. Resolution of all acute toxic effects of prior anticancer therapy to grade ≤ 1 as determined by the NCI-CTCAE v.5.0 criteria (except for alopecia or other toxicities not considered a safety risk for the patient at Investigator's discretion).
14. For women of childbearing potential who are sexually active with a non-sterilized male partner: must have a negative serum pregnancy test within 14 days before study treatment initiation. In addition, agreement to remain abstinent (refrain from heterosexual intercourse) or use one highly effective method of birth control or two effective contraceptive methods, as defined in the protocol from the time of screening until 7 months after the last dose of study treatments. Female patients must agree to refrain from egg cell donation and breastfeeding during this same period.
15. Male participants who intend to be sexually active with a female partner of childbearing potential must be surgically sterile or use highly effective contraceptive methods, or two effective contraceptive methods, as defined in the protocol from the time of screening until 4 months after the last dose of T-DXd or 7 months after the last dose of PHESGO to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same period. Not engaging in heterosexual activity (sexual abstinence) for the duration of the study and drug washout period is an acceptable practice if this is the preferred usual lifestyle of the participant the last dose of study treatments.
16. Patient must be accessible for treatment and follow-up.

Exclusion Criteria:

An individual who meets ANY of the following criteria will be excluded from participation in this trial:

1. Current participation in another therapeutic clinical trial, except other translational studies.
2. Treatment with approved or investigational cancer therapy within 14 days prior to initiation of study drugs.
3. Has previously been treated with T-DXd in the adjuvant or neoadjuvant setting.
4. Known active uncontrolled or symptomatic central nervous system (CNS) metastases and/or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth.

   Note: Patients with a history of CNS metastases are eligible if they have been previously treated with local therapy, are clinically stable, and off anticonvulsants and steroids for at least 14 days before the first dose of study treatment.
5. Concurrent malignancy or malignancy within 5 years of study enrollment with the exception of carcinoma in situ of the cervix, non-melanoma skin carcinoma, or stage I uterine cancer. For other cancers considered to have a low risk of recurrence, discussion with the Sponsor's Medical Monitor is required.
6. Known allergy or hypersensitivity reaction to any investigational medicinal products (IMPs) or their incorporated substances.
7. Palliative radiotherapy with a limited field of radiation within 2 weeks or with wide field of radiation or to more than 30% of the bone marrow within 4 weeks prior to start of study treatment.
8. Major surgical procedure or significant traumatic injury within 14 days before the first dose of study treatment or anticipation of need for major surgery within the course of the study treatment.
9. Has an active cardiac disease or a history of cardiac dysfunction or severe conduction abnormalities including, but not confined, to any of the following:

   1. Unstable angina pectoris, documented myocardial infarction, or symptomatic cardiac heart failure (CHF) (New York Heart Association [NYHA] Class II-IV) within six months prior to study entry.
   2. Poorly controlled hypertension (i.e., systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg).
   3. Symptomatic pericarditis.
   4. Left ventricular ejection fraction (LVEF) < 55 % as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO).
   5. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, or ventricular tachycardia), which is symptomatic or requires treatment (NCI-CTCAE grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, asymptomatic sustained ventricular tachycardia, or higher-grade atrioventricular [AV]-block, such as second-degree AV-block Type 2 [Mobitz 2] or third-degree AV-block). Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers will be permitted to enroll.
   6. QT Interval Corrected by Fridericia's formula (QTcF) prolongation to > 470 ms (females) or > 450 ms (males) based on average of the screening triplicate 12-lead ECG.
   7. History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
   8. Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
10. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (e.g., pulmonary emboli within three months of the study enrolment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, post COVID-19 pulmonary fibrosis, etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or prior pneumonectomy.
11. Has a history of non-infectious interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
12. Pregnant or lactating women or patients not willing to apply highly effective contraception as defined in the protocol.
13. Current known infection with hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients with past HBV infection or resolved HBV infection (defined as having a negative hepatitis B surface antibody [HBsAg] test and a positive hepatitis B core antibody [HBcAb] test, accompanied by a negative HBV DNA test) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
14. Has active primary immunodeficiency, known human immunodeficiency virus (HIV) infection.
15. Other active uncontrolled infection at the time of enrollment.
16. Receipt of live or attenuated vaccine within 30 days prior to the first dose of study treatment.
17. A history of uncontrolled seizures, CNS disorders or serious and/or unstable pre-existing psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs or interfering with subject safety.
18. Has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate patient participation in the clinical study.
19. Known substance abuse or any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation.
20. Inability or unwillingness to comply with study and follow-up procedures in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
1-year PFS rate | Baseline up to 12 months
  To determine the rate of patients with absence of disease progression or death from any cause at 1 year after the treatment initiation with T-DXd followed by PHESGO, as determined locally by the investigator using RECIST v.1.1
3-year OS rate | Through study completion, an average of 36 months
  To determine the rate of patients alive at 3 years after treatment initiation with T-DXd followed by PHESGO.

SECONDARY OUTCOMES:
Global PFS rate | Through study completion, an average of 36 months
  To assess the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of PFS, defined as the period from treatment initiation until to the first occurrence of disease progression as determined locally by the investigator assessment using RECIST v.1.1 or death from any cause, whichever occurs first.
Global OS rate | Through study completion, an average of 36 months
  To assess the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of OS, defined as the period from treatment initiation to death from any cause, as determined locally by the investigator.
Objective response rate (ORR) | Through study completion, an average of 36 months
  To determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of ORR, defined as the rate of patients with complete response (CR) or partial response (PR), as determined locally by the investigator using RECIST v.1.1.
Clinical benefit rate (CBR) | Through study completion, an average of 36 months
  To determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of CBR, defined as the rate of patients with objective response (CR or PR), or stable disease for at least 24 weeks, as determined locally by the investigator using RECIST v.1.1.
Time to response (TTR) | Through study completion, an average of 36 months
  To determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of TTR, defined as the period from treatment initiation to the first objective tumor response (tumor shrinkage of ≥ 30%) observed for patients who achieved a CR or PR, as determined locally by the investigator using RECIST v.1.1.
Duration of response (DoR) | Through study completion, an average of 36 months
  To determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of DoR, defined as the period from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using RECIST v.1.1.
Best percentage of change | Through study completion, an average of 36 months
  To determine the efficacy of induction treatment with T-DXd followed by PHESGO as maintenance therapy in terms of best percentage of change from baseline in the size of target tumor lesions, defined as the biggest decrease, or smallest increase if no decrease will be observed, as determined locally by the investigator using RECIST v.1.1.
Quality of life (QoL) | Baseline up to 42 weeks
  To evaluate changes during induction treatment with T-DXd and maintenance therapy with PHESGO in terms of patient-reported outcome (PRO) assessments of QoL and treatment-related symptoms as measured by selected scales from the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients questionnaire (QLQ-C30) and breast cancer module (QLQ-BR45), and from the EuroQol Group 5-level EQ-5D version (EQ-5D-5L) questionnaire.
Safety and tolerability | Through study completion, an average of 36 months
  To evaluate the safety and toxicity profile of treatment with T-DXd followed by PHESGO in all patients as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

OTHER OUTCOMES:
Efficacy endpoints according to protein expression status on baseline tissue samples | Through study completion, an average of 36 months
  To determine the protein expression status (IHC and proteomics on baseline tissue samples and its potential correlation with treatment efficacy endpoints.
Efficacy endpoints according to circulating tumor DNA (ctDNA) level changes in blood samples | Through study completion, an average of 36 months
  To assess the association of treatment efficacy endpoints with ctDNA level changes between liquid biopsy samples obtained at baseline and at different timepoints during the treatment period, and at the end of treatment.
Efficacy endpoints according to mutational profiling on baseline tissue samples | Through study completion, an average of 36 months
  To determine mutational profiling on baseline tissue samples and its relationship with efficacy endpoints.
Efficacy endpoints according to gene expression profiling on baseline tumor samples | Through study completion, an average of 36 months
  To evaluate the potential correlation of gene expression profiling on baseline tumor samples with the disease status or patient outcomes.
Efficacy endpoints according to clinicopathological characteristics | Through study completion, an average of 36 months
  To determine the relationship between different clinicopathological characteristics and efficacy endpoints.
Efficacy endpoints according to medical imaging biomarkers | Through study completion, an average of 36 months
  To determine new oncological biomarkers of radiological imaging - such as growth rate of tumor derived by tumor growth rate modeling or tumor heterogeneity according to quantitative estimation through radiomics - that could help to better understand the efficacy of drug treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Cortés, MD, PhD, Principal Investigator — Institute of Breast Cancer, Quirón Group, Barcelona (Spain); Antonio Llombart-Cussac, MD, Principal Investigator — Arnau de Vilanova Hospital, Valencia (Spain); José M Pérez-García, MD, Principal Investigator — International Breast Cancer Center (Spain)
Locations (36):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Northwell Health, New York, New York
- France (3):
  - Institute Paoli Calmettes, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Tenon AP-HP, Paris
- Germany (4):
  - Marienhospital Bottrop GmbH Klinik für Gynäkologie und Geburtshilfe, Bottrop
  - Kliniken Essen Mitte, Essen
  - Mammazentrum HH, Hamburg
  - Klinikum der Universität München, München
- Italy (4):
  - Humanitas Gavazzeni, Bergamo
  - Instituto Europeo di Oncologia, Milan
  - University Hospital Maggiore della Carita, Novara
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Spain (23):
  - Hospital del Vinalopó, Alicante
  - Hospital General Universitario Dr. Balmis (Alicante), Alicante
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Institut Català d' Oncologia L'Hospitalet (ICO), Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Clínico San Cecilio de Granada, Granada
  - Hospital Universitario de León, León
  - Hospital Beata María Ana, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Quirónsalud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Instituto Valenciano de Oncología (IVO), Valencia